CLINICAL TRIAL: NCT02158871
Title: Beyond Silence: Comparing the Impact of Contact-based Education With Mental Health Literacy Training on Early Intervention for Healthcare Workers With Mental Health Issues
Brief Title: Impact Study of Workplace Mental Health Education on Early Intervention for Healthcare Workers With Mental Health Issues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Ontario Mental Health Foundation (Other Government); Hamilton Health Sciences Corporation (Other); St. Joseph's Health Care London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MBSi14-385
Record Dates: First submitted 2014-05-29; First posted 2014-06-09 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Mental Health Impairment
Keywords: Education; Early intervention; Workplace; Stigma; Mental Health Literacy
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contact-based mental health education (Experimental): The "Beyond Silence' program is 12 hours in length: six 1.5-2 hour in-person group sessions every other week, plus five online sessions between each of the in-person sessions.
  Interventions: Behavioral: Beyond Silence
- Mental health literacy training (Active Comparator): "Mental Health First Aid" training consists of twelve hours of standardized, module-based mental health literacy training offered in a group format. It will be offered as 2 full-day training sessions (or four half-day sessions).
  Interventions: Behavioral: Mental Health First Aid (MHFA)

INTERVENTIONS:
Behavioral: Beyond Silence — Pilot data from initial phases of the project and best practice principles in contact based education and adult learning theory informed curriculum design. The six in-person sessions use workplace-based vignettes to prompt reflection and discussion, build mental health literacy, reduce stigma, and promote communication and coping skill development. The virtual sessions use a secure online discussion board for participants to explore relevant online resources. All sessions will be co-led by trained peer educators; employees who have personally experienced mental ill health and recovery and are viewed as credible leaders within the organization. They will be recruited and trained to effectively teach the content, share personal experiences, and facilitate discussion.
  Other Names: Contact-based mental health education
  Arms: Contact-based mental health education
Behavioral: Mental Health First Aid (MHFA) — MHFA is a standardized, twelve-hour educational program designed to teach participants how to recognize the early warning signs of mental illness, how to provide initial help to someone in a mental health crisis, and how to support people who are developing mental health problems. It is an evidence-based approach that originated in Australia, but is being implemented across Canada, under the leadership of the Mental Health Commission of Canada. Leadership of the MHFA will be provided by an employee in each organization who has been trained through the 5-day national MHFA instructor training program. The instructor does not share any personal experiences regarding mental health issues.
  Other Names: Mental health literacy training
  Arms: Mental health literacy training

SUMMARY:
The purpose of this study is to compare the impact of a new workplace-based mental health peer education program with standardized mental health literacy training on early intervention and support for healthcare employees with mental health issues. Participants are healthcare workers who volunteer to participate in one of the two twelve-hour group education programs. It is hypothesized that the customized "Beyond Silence" peer education program led by trained staff members with personal experience of mental ill-health will be more effective in reducing the stigma associated with help-seeking and help-outreach regarding mental ill-health in the workplace. The comparison group is a standardized mental health literacy training program that has been widely implemented in both Canada and around the world. Change in help-seeking/help-outreach behavior, mental health knowledge and beliefs of participants will be assessed at three-month intervals; before, after and three months following the educational intervention.

DETAILED DESCRIPTION:
The target sample of 200 employee participants will be recruited from two healthcare organizations. The Beyond Silence program is based on principles of contact-based education, and will include six 1.5-2 hour in-person sessions conducted every other week, interspersed with five online resource sessions. The Mental Health First Aid training is a standardized, 12-hour evidence-based mental health literacy training program that has been implemented in a range of national and international settings. This program is typically offered over two full days.

ELIGIBILITY:
Inclusion Criteria:

* Employee (full-time, part-time or contract) in the participating healthcare organization
* Willing and able to participate in 12 hours of training outside of paid work hours
* Able to understand and speak English

Exclusion Criteria:

* Prior training in either of the two educational approaches

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in help-seeking behavior | Baseline, post-intervention, 3 month follow-up
  Participants will be asked to report whether they accessed any services from a list of 10 health, workplace and community service options. Questions regarding service utilization are adapted from the 2012/2012 Canadian Community Health survey, in order to provide a population reference, plus several work-related services (eg. EAP, union) are added as an option. Participants may endorse more than one of the behaviors, and a summative score of the number of behaviors will be used to measure change in help-seeking.
Change from baseline in help-outreach behavior | Baseline, post-intervention, 3 month follow-up
  Self-report of personal contact with a co-worker about mental health problems (yes/no), and any contact over the past 6 months (yes/no). If contact did occur, participants will be asked whether they provided help to the co-worker, and if so, to identify the type of help from a list of 10 possible options. The list of "outreach" behaviors was based on Mental Health First Aid program evaluation (e.g. 'spent time listening to problem', 'recommend professional help'), with an adaptation to include a several work-specific options (e.g., 'recommend EAP', 'offered assistance with job duties'). Participants are invited to check all behaviors that apply (with an open-ended option), and scoring is based on one point per action, with a summative score used to track change. In addition to the behavior list, participants will be asked to rate their confidence in providing help on a 7 point Likert scale.

SECONDARY OUTCOMES:
Change from baseline in degree of stigma towards co-workers with a mental illness | Baseline, post-intervention, 3 month follow-up
  The Mental Health Commission of Canada Opening Minds Scale for Healthcare Providers will be used; a 20-item questionnaire designed to evaluate the attitudes of healthcare providers towards people with mental illness. The tool has good internal consistency (α=.82), and satisfactory test-retest reliability (ICC=.66), with limited impact of social desirability.
Change from baseline in mental health literacy | Baseline, post-intervention, 3 month follow-up
  Four vignettes of employees with workplace mental health issues will be used to assess awareness of issues and when/how to respond to these issues in the workplace. The vignettes are adapted for a healthcare workplace based on a review of vignettes reported in the literature, as well as analysis of key issues reported in the pilot phase of the study. Vignettes will incorporate differences in gender, nature and severity of illness, and a 7 point Likert scale from novice to expert will be used to track key dimensions of literacy, including perceived knowledge about the condition, what to say/do and what resources to access.
Change from baseline in attitudes toward professional help-seeking for mental health issues | Baseline, post-intervention, 3 month follow-up
  The Attitudes Toward Seeking Professional Psychological Help Scale-short form (ATSPPHS), a 10 question survey using a four point Likert-type scale response will be used to track beliefs and intent to seek professional help. It is a widely used scale with good internal consistency (α=.78), and criterion validity supported by links between scale scores and mental healthcare use.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra E Moll, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario

REFERENCES:
- [Derived] Richardson R, Dale HE, Robertson L, Meader N, Wellby G, McMillan D, Churchill R. Mental Health First Aid as a tool for improving mental health and well-being. Cochrane Database Syst Rev. 2023 Aug 22;8(8):CD013127. doi: 10.1002/14651858.CD013127.pub2. PMID 37606172
- [Derived] Moll S, Patten SB, Stuart H, Kirsh B, MacDermid JC. Beyond silence: protocol for a randomized parallel-group trial comparing two approaches to workplace mental health education for healthcare employees. BMC Med Educ. 2015 Apr 16;15:78. doi: 10.1186/s12909-015-0363-9. PMID 25880303